CLINICAL TRIAL: NCT00776321
Title: A Placebo Controlled, Double Blind, Randomised, 12-Week, Phase ii Study to Assess the Safety and Efficacy of KB2115 in Patients With Primary Hypercholesterolemia
Brief Title: Eprotirome for the Treatment of Dyslipidemia, Efficacy and Safety 12-Week, Phase ii Study to Assess the Safety and Efficacy of KB2115 in Patients With Primary Hypercholesterolemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karo Bio AB (Industry)
Responsible Party: Jens Kristensen, MD PhD, Chief Medical Officer, Karo Bio AB
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EudraCT No: 2006-003191-35
Record Dates: First submitted 2008-10-17; First posted 2008-10-21 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Primary Hypercholesterolemia
Keywords: hypercholesterolemia; dyslipidemia; thyroid; safety
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias; Thyroid Diseases | interventions — 3-((3,5-dibromo-4-(4-hydroxy-3-(1-methylethyl)phenoxy)phenyl)amino)-3-oxopropanoic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- Eprotirome dose 1 (Experimental)
  Interventions: Drug: Eprotirome
- Eprotirome dose 2 (Experimental)
  Interventions: Drug: Eprotirome

INTERVENTIONS:
Drug: Eprotirome
  Other Names: KB2115
  Arms: Eprotirome dose 1; Eprotirome dose 2
Drug: Placebo
  Arms: 1

SUMMARY:
Eprotirome (KB2115) is a liver selective thyroid hormone that can induce hyperthyroidism in the liver, while an euthyroid state is preserved in the extrahepatic tissue. Eprotirome has in a clinical 2-weeks studies demonstrated pronounced reduction of independent risk factors for the development of atherosclerotic cardiovascular diseases.

The purpose of the study is to assess the efficacy and safety of KB2115 as monotherapy following 12 weeks of exposure compared to placebo. The aim of the study is to assess efficacy (LDL-cholesterol lowering effects) and safety of KB2115.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of hypercholesterolemia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2006-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
LDL cholesterol | Week 12

SECONDARY OUTCOMES:
Lipid variables, Thyroid hormone levels, Bone markers,DEXA, ECG, Echocardiography, liver enzymes | 12 week

CONTACTS AND LOCATIONS:
Locations (1):
- Jens Kristensen, Huddinge, Sweden